CLINICAL TRIAL: NCT03900572
Title: A Randomized, Double-Blind and Placebo-Controlled Phase I Study to Evaluate the Safety and Immunogenicity of a 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 and 58) Recombinant Vaccine (Pichia Pastoris) in 9 to 45 Year Old Chinese Females
Brief Title: A Study of Safety and Primary Immunogenicity of 9-valent HPV Recombinant Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Zerun Biotechnology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 312-HPV-2001
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: HPV Infections
Keywords: Human Papilloma Virus; Papillomavirus vaccines; Cervical Cancer; Genital Warts
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Condylomata Acuminata | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV vaccine (Experimental): Subjects receive 3 doses of 9-valent HPV vaccine according to a 0, 2, 6-month schedule.
  Interventions: Biological: HPV Vaccine
- Placebo (Placebo Comparator): Subjects received 3 doses of Placebo according to a 0, 2, 6-month schedule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: HPV Vaccine — Intramuscular injection, 3 doses
  Arms: HPV vaccine
Drug: Placebo — Intramuscular injection, 3 doses
  Arms: Placebo

SUMMARY:
A randomized, double-blind and placebo-controlled phase I study to evaluate the safety and immunogenicity of a 9-valent Human Papillomavirus (HPV) vaccine, administered intramuscularly according to a 0, 2, 6-month schedule in 9 to 45 years old healthy Chinese females.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females, 9 to 45 years old (inclusive).
* 9 to 17 years old participants: able to prove their identities and provide their legal guardians' identity information.
* Legal guardians of the 9 to 17 years old participants: able to understand (not illiterate) and agree to co-sign the informed consent forms with participants
* 18 to 45 years old participants: able to prove their legal identities.
* 18 to 45 years old participants: able to understand (not illiterate) the study and agree to sign the informed consent form.
* Child bearing age participants: agree not to become pregnant by using proper contraception means in the 7-month study period.

Exclusion Criteria:

* History of cervical cancer or genital warts.
* History HPV vaccination or history of participation in HPV vaccine trial.
* History of severe allergy which needs medical intervention such as swelling of the mouth and throat, difficulty breathing, hypotension or shock.
* Skin abnormality at injection site including inflammation, sclerosis, redness, swelling, and extensive scars.
* History of allergy to vaccine or vaccine components including aluminum phosphate, histidine and Polysorbate 80, and severe adverse reactions in past vaccination.
* Medical history of epilepsy, convulsions, seizures , or family history of mental illness.
* Medical conditions including immunocompromised or diagnosed as congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease or other autoimmune diseases and received immunosuppressants in 6 months prior to first vaccination.
* History of asthma, thyroidectomy, angioneurotic edema, diabetes, and malignancy.
* Asplenia, functional asplenia, or any circumstances as a result of asplenia or splenectomy
* Diagnosis as coagulation abnormalities such as clotting factor deficiency, platelet abnormalities or having significant bruising, or coagulation disorder
* Being diagnosed with acute illnesses or acute onset of chronic illness during the last 3 days.
* Treatment with immunoglobulins or other blood-derived products within 3 months prior to Day 0 vaccination.
* Having received subunit or inactivated vaccine within 14 days prior to Day 0 vaccination or received attenuated vaccine within 28 days prior to Day 0 vaccination.
* Fever before vaccine administration with axillary temperature higher than 37.0°C.
* Currently breastfeeding, and being pregnant including pregnancy test positive.
* History of hypertension: Participants of 13 to 45 years of age have their respective systolic blood pressure greater than 150 mmHg and/or diastolic blood pressure greater than 100 mmHg; or participants of 9 to 12 years of age demonstrate their respective systolic blood pressure higher than 120 mmHg and/or diastolic blood pressure higher than 80 mmHg.
* Exhibits of abnormal lab test parameters.
* Any other factors which might affect any individual to be enrolled in the study according to the investigator's judgment.

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects Reporting Solicited Local Symptoms | During a 8-day period (Day 0-7) following each vaccination
  Solicited local symptoms assessed including pain, redness, swelling, induration and itching.
Percentage of Subjects Reporting Solicited General Symptoms | During a 8-day period (Day 0-7) following each vaccination
  Solicited general symptoms assessed including fever, headache, fatigue, nausea, diarrhea, vomiting, myalgia, allergic reaction
Percentage of Subjects Reporting Unsolicited Adverse Events (AEs) | Within 31 days (Day 0-30) after any vaccination
  An unsolicited adverse event is defined as any adverse event (AE) reported in addition to those solicited during the clinical study.
Percentage of Subjects Reporting Serious Adverse Events (SAE) | Throughout the study period (up to Month 12)
  Serious adverse events are defined as medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.

SECONDARY OUTCOMES:
Seroconversion Percentages to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 | 30 days after the third dose (Month 7)
  Seroconversion is defined as a participant who was anti-HPV seronegative at Day 0 (before vaccination) and became seropositive 30days after the third dose (Month 7).
Geometric Mean Titers (GMT) of HPV serotype-specific antibody | 30 days after the third dose (Month 7)
  HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 specific antibodies GMT

CONTACTS AND LOCATIONS:
Overall Officials: Xuecheng LIU, BS, Principal Investigator — Sichuan Provincial Center for Disease Prevention and Control
Locations (1):
- Sichuan Provincial Center for Disease Prevention and Control, Chengdu, Sichuan, China